CLINICAL TRIAL: NCT03008161
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Multiple Dose, Dose Escalation Study of NPT088 in Patients With Probable Alzheimer's Disease
Brief Title: Multiple Dose Safety Study of NPT088 in Patients With Mild to Moderate Probable Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Proclara Biosciences, Inc. (Industry)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPT088-CL002
Record Dates: First submitted 2016-12-23; First posted 2017-01-02 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Alzheimer Disease
Keywords: GAIM; amyloid; anti-aBeta; anti-tau
MeSH Terms: conditions — Alzheimer Disease | interventions — Immunoglobulin G

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): Participants will receive monthly IV infusions of either low dose NPT088 (6 participants) or placebo (3 participants) for a total of 6 months
  Interventions: Drug: NPT088; Drug: Placebo
- Cohort 2 (Experimental): Participants will receive monthly IV infusions of either mid-low dose NPT088 (6 participants) or placebo (3 participants) for a total of 6 months
  Interventions: Drug: NPT088; Drug: Placebo
- Cohort 3 (Experimental): Participants will receive monthly IV infusions of either mid-high dose NPT088 (16 participants) or placebo (8 participants) for a total of 6 months
  Interventions: Drug: NPT088; Drug: Placebo
- Cohort 4 (Experimental): Participants will receive monthly IV infusions of either high dose NPT088 (16 participants) or placebo (8 participants) for a total of 6 months
  Interventions: Drug: NPT088; Drug: Placebo

INTERVENTIONS:
Drug: NPT088 — IgG1 Fc-GAIM fusion protein, a recombinant fusion protein
  Other Names: IgG1; fusion protein; GAIM; anti-Abeta; anti-Tau
Drug: Placebo — Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of multiple doses of NPT088 in patients with mild to moderate probable Alzheimer's Disease. The study will also evaluate the pharmacokinetics, immunogenicity and exploratory pharmacodynamic characteristics of multiple doses of NPT088.

DETAILED DESCRIPTION:
This study is a multicenter Phase 1, randomized, double-blind, placebo-controlled, multiple-dose, dose-escalation safety and tolerability study of NPT088 or placebo in patients with Probable AD with a MMSE score of 16-27. Enrolled patients will receive an intravenous infusion of NPT088 or placebo once a month for six months during this study. Four dose cohorts are planned with the first two cohorts enrolling 9 patients each (6 NPT088: 3 placebo) and the final two cohorts enrolling 24 patients each (16 NPT088: 8 placebo) for a total of 66 patients (44 NPT088: 22 placebo).

ELIGIBILITY:
Inclusion Criteria: For enrollment in the study, participants must

* be between 50 and 85 years of age, inclusive
* have a Mini Mental State Examination (MMSE) scores between 16-27 (inclusive)
* have a Modified Hachinski Score of less than or equal to 4
* have a diagnosis of Probable Alzheimer's Disease (AD) according to consensus criteria defined by the National Institute on Aging-Alzheimer's Association work group
* have a Clinical Dementia Rating Scale (CDR) of 0.5 or 1.0, with the memory box score equal to or greater than 0.5
* have a positive florbetapir positron emission tomography (PET) amyloid scan
* consent to apolipoprotein E (ApoE) genotyping
* be willing to undergo repeat Magnetic Resonance Imaging (MRI) and PET imaging
* be on stable doses of allowed medications for at least 30 days prior to Screening. Concurrent treatment with cholinesterase inhibitors and/or memantine is allowed
* be in good healthy apart from the clinical diagnosis of AD
* have a dedicated Caregiver who provides care at least 4 hours a day for 4 days a week and will provide informed consent for their participation

Exclusion Criteria: For enrollment in the study, participants must NOT:

* have a history of, or screening MRI indicative of any significant brain abnormality
* have any major medical illness or unstable medical condition or in the opinion of the Investigator have any reason that may interfere with the participants ability to comply with the study procedures and abide by study restrictions or with the ability to interpret safety data
* reside in a nursing home or need 24-hour care and supervision
* take excluded medications
* have exclusionary values on the Screening blood and urine sample
* have been treated with immunomodulators to treat AD
* have participated in an investigational drug or device study within 90 days
* have a known allergy to study drug

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Baseline to Week 32

SECONDARY OUTCOMES:
Multiple dose pharmacokinetic (PK) serum concentrations of NPT088 | Up to Week 32
Multiple dose PK CSF concentrations of NPT088 | Up to Week 32
Multiple dose immunogenicity of NPT088 | Up to Week 32

OTHER OUTCOMES:
Change from baseline in florbetapir-fluorine-18 positron emission tomography (PET) imaging in certain brain areas | Baseline and Week 24
Change from baseline in [18F] MNI-960 PET imaging in certain brain areas | Baseline and Week 24
Change in CSF or blood biomarkers | Up to Week 32

CONTACTS AND LOCATIONS:
Overall Officials: Proclara Biosciences, Study Director — Proclara
Locations (23):
- United States (23):
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Neurology Center of North Orange County, Fullerton, California
  - Collaborative Neuroscience Network, Long Beach, California
  - Southern California Research, Simi Valley, California
  - Associated Neurologists of Southern Connecticut, Fairfield, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Compass Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Axiom Clinical Research, Tampa, Florida
  - Compass-The Villages, The Villages, Florida
  - Medical Research and Health Education Foundation, Columbus, Georgia
  - NeuroStudies LLC, Decatur, Georgia
  - Princeton Medical Institute, Princeton, New Jersey
  - Neurological Associates of Albany, Albany, New York
  - Integrative Clinical Trials, Inc., Brooklyn, New York
  - Alzheimer's Memory Center, Charlotte, North Carolina
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Abington Neurological Associates, Ltd, Willow Grove, Pennsylvania
  - Neurology Clinic, PC, Cordova, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krishnan R, Tsubery H, Proschitsky MY, Asp E, Lulu M, Gilead S, Gartner M, Waltho JP, Davis PJ, Hounslow AM, Kirschner DA, Inouye H, Myszka DG, Wright J, Solomon B, Fisher RA. A bacteriophage capsid protein provides a general amyloid interaction motif (GAIM) that binds and remodels misfolded protein assemblies. J Mol Biol. 2014 Jun 26;426(13):2500-19. doi: 10.1016/j.jmb.2014.04.015. Epub 2014 Apr 22. PMID 24768993
- [Background] Levenson JM, Schroeter S, Carroll JC, Cullen V, Asp E, Proschitsky M, Chung CH, Gilead S, Nadeem M, Dodiya HB, Shoaga S, Mufson EJ, Tsubery H, Krishnan R, Wright J, Solomon B, Fisher R, Gannon KS. NPT088 reduces both amyloid-beta and tau pathologies in transgenic mice. Alzheimers Dement (N Y). 2016 Jul 14;2(3):141-155. doi: 10.1016/j.trci.2016.06.004. eCollection 2016 Sep. PMID 29067301
- [Background] Krishnan R, Hefti F, Tsubery H, Lulu M, Proschitsky M, Fisher R. Conformation as the Therapeutic Target for Neurodegenerative Diseases. Curr Alzheimer Res. 2017;14(4):393-402. doi: 10.2174/1567205014666170116152622. PMID 28093972